CLINICAL TRIAL: NCT05034783
Title: A Pilot Prospective Comparison of [68Ga]Ga-HBED-CC-exendin-4 and [68Ga]Ga-NOTA-exendin-4 PET/CT Imaging in the Same Group of Insulinoma Patients
Brief Title: [68Ga]Ga-HBED-CC-exendin-4 and [68Ga]Ga-NOTA-exendin-4 PET/CT Imaging in the Same Group of Insulinoma Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-NM-EX4
Record Dates: First submitted 2021-09-02; First posted 2021-09-05 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Insulinoma
MeSH Terms: conditions — Insulinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [68Ga]Ga-HBED-CC-exendin-4 and [68Ga]Ga-NOTA-exendin-4 PET/ CT scan (Experimental): Patients of Insulinoma PET/CT imaging: In two consecutive days each patient underwent a 60-min dynamic PET/CT scan after intravenous administration of [68Ga]Ga-HBED-CC-exendin-4 and [68Ga]Ga-NOTA-exendin-4, respectively.
  Interventions: Drug: [68Ga]Ga-HBED-CC-exendin-4; Drug: [68Ga]Ga-NOTA-exendin-4

INTERVENTIONS:
Drug: [68Ga]Ga-HBED-CC-exendin-4 — Intravenous injection of one dosage of 74-111 MBq (2-3 mCi) [68Ga]Ga-HBED-CC-exendin-4. Tracer doses of [68Ga]Ga-HBED-CC-exendin-4 will be used to image lesions of insulinoma by PET/CT.
  Other Names: [68Ga]Ga-HBED-CC-exendin-4 injection
Drug: [68Ga]Ga-NOTA-exendin-4 — Intravenous injection of one dosage of 74-111 MBq (2-3 mCi) [68Ga]Ga-NOTA-exendin-4. Tracer doses of [68Ga]Ga-NOTA-exendin-4 will be used to image lesions of insulinoma by PET/CT.
  Other Names: [68Ga]Ga-NOTA-exendin-4 injection

SUMMARY:
Glucagon-like peptide-1 receptor (GLP-1R)-targeted PET imaging with 68Ga-labeled compounds is able to provide superior sensitivity and specificity to detect insulinoma, like the widely studied [68Ga]Ga-NOTA-exendin-4. This pilot study was prospectively designed to evaluate the early dynamic distribution of [68Ga]Ga-HBED-CC-exendin-4, a novel radiopharmaceutical targeting GLP-1R, which was compared with [68Ga]Ga-NOTA-exendin-4 in the same group of insulinoma patients.

DETAILED DESCRIPTION:
Insulinoma is the most common cause of endogenous hyperinsulinemic hypoglycemia in adult patients without diabetes. The only curative treatment of an insulinoma is its surgical removal. Therefore, exact preoperative localization of the insulinoma is critical to planning the surgical intervention. MR imaging, CT, or endoscopic ultrasound is normally used to localize insulinomas. However, the small size of the tumors (often,1 cm) limits the sensitivity of these methods. In recent years, a new receptor-targeted imaging technique, glucagon-like peptide-1 receptor (GLP-1R) imaging, for detecting insulinoma has been established. GLP-1R is expressed on benign insulinoma cell surfaces with very high incidence (>90%) and density (8,133 dpm/mg of tissue). No other peptide receptor has been found to exhibit such high expression levels in insulinoma. [68Ga]Ga-HBED-CC-exendin-4, a novel radiopharmaceutical targeting GLP-1R, with the urea fragment of a conjugate that employs the HBED-CC chelator for labeling with 68Ga in order to In order to reduce the accumulation of radioactivity in the kidneys. This pilot study was prospectively designed to evaluate the early dynamic distribution of [68Ga]Ga-HBED-CC-exendin-4 compared with [68Ga]Ga-NOTA-exendin-4 in the same group of Insulinoma patients.

ELIGIBILITY:
Inclusion Criteria:

* confirmed treated or untreated insulinoma patients;
* [68Ga]Ga-HBED-CC-exendin-4 and [68Ga]Ga-NOTA-exendin-4 PET/CT within two consecutive days;
* signed written consent.

Exclusion Criteria:

* pregnancy;
* breastfeeding;
* known allergy against exendin-4;
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Metabolic parameters | through study completion, an average of 1 year
  the early dynamic distribution (SUVmax in tumor lesions and SUVmean in normal organs at different time points) of [68Ga]Ga-HBED-CC-exendin-4 in comparison with [68Ga]Ga-NOTA-exendin-4 in the same group of insulinoma patients.

SECONDARY OUTCOMES:
Diagnostic value | through study completion, an average of 1 year
  Sensitivity and Specificity of [68Ga]Ga-HBED-CC-exendin-4 for insulinoma in comparison with [68Ga]Ga-NOTA-exendin-4 PET/CT.

OTHER OUTCOMES:
GLP-1R expression and SUV | through study completion, an average of 1 year
  Correlation between GLP-1R expression and SUV in PET

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li L, Wang G, Wang J, Ma H, Chen J, Wang R, Pan Q, Hong H, Jin W, Kung HF, Zhu L, Luo Y, Zhu Z. Glucagon-Like Peptide-1 Receptor-Targeted PET/CT With 68 Ga-HBED-CC-Exendin-4 in Localizing Insulinoma : A Head-to-Head Comparison to 68 Ga-NOTA-Exendin-4. Clin Nucl Med. 2025 Jan 1;50(1):38-43. doi: 10.1097/RLU.0000000000005533. Epub 2024 Nov 8. PMID 39499011